CLINICAL TRIAL: NCT06491836
Title: The Effect of an Oligoantigenic Diet on Core Symptomatology of Children With Attention-Deficit /Hyperactivity Disorder (ADHD).
Brief Title: Oligoantigenic Diet and Core Symptomatology of Children With Attention-Deficit /Hyperactivity Disorder (ADHD).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Haya Essam Ibrahim, lecturer of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MS157/2024
Record Dates: First submitted 2024-06-28; First posted 2024-07-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Patients who will follow food regimen without any food restriction. (Active Comparator)
  Interventions: Other: Food regimen without food restrictions.
- Arm 2: Patients who will follow food regimen based on oligoantigenic diet. (Experimental)
  Interventions: Dietary Supplement: oligoantigenic diet

INTERVENTIONS:
Dietary Supplement: oligoantigenic diet — Oligoantigenic diet that will cover recommended daily allowance (RDA) of macronutrients and micronutrients according patients' ages according to our available sources of food in our culture and the diet consists typically of meat (e.g. chicken and lamb), carbohydrate sources (e.g., potatoes and rice), fruits (e.g., bananas, pears and apples), vegetables (e.g., cucumbers, carrot, lettuce, cauliflower, turnips, cabbage and broccoli)
  Arms: Arm 2: Patients who will follow food regimen based on oligoantigenic diet.
Other: Food regimen without food restrictions. — Food regimen that will cover recommended daily allowance (RDA) for macronutrients and micronutrients according patients' ages without any food restriction
  Arms: Arm 1: Patients who will follow food regimen without any food restriction.

SUMMARY:
Fifty patients who diagnosed as ADHD syndrome according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) Criteria aged from 6 to 16 years old will be assigned randomly into 2 arms: arm 1: the patients will follow food regimen that cover recommended daily allowance (RDA) for macronutrients and micronutrients suitable for their ages without any food restriction, arm 2: the patients will follow food regimen that cover (RDA) for macronutrients and micronutrients suitable for their ages based on Oligoantigenic diet (OAD). Psychiatric assessment will be done before intervention and after 3 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children fulfilled DSM (5) Criteria for ADHD syndrome aged from 6 to 16 years old on stable pharmacotherapy 8 weeks prior to enrollment with intention to maintain ongoing therapies constant throughout the trial.

Exclusion Criteria:

* Presence of other medical conditions as chronic medical illness or other neuropsychiatric disorders
* Intelligence quotient (IQ) of patients less than 80%.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Conner's Parent Rating Scales-Revised (CRS-R) | 3 months
  This tool is used to assess the profile and severity of symptoms, response to treatment and follow up studies. Items will be scored on 14 subscales of symptoms including opposition, cognitive problems, inattention and hyperactivity. It is usually considered normal when T-scores are less than 60, while scores above 60 are signs of academic, behavioral or social issues.
Child Behavior Checklist (CBCL/6-18) | 3 months
  It is designed to obtain parents'/caregivers' reports of their children's problems and it is a reliable tool for assessing the traits associated with childhood mental health issues.
The Continuous Performance Test (CPT) | 3 months
  It is a measurement of sustained attention deficits. It requires participants to respond to predesignated targets among stimuli that will be presented at a rapid fixed rate.
Clinical Global Impression | 3 months
  Scale is designed to assess the effectiveness of a particular treatment: CGI-severity scale (CGI-S) assessing illness severity and CGI-C assessing global improvement or change. CGI-S will measure illness severity at baseline and after treatment on a scale of seven points

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided